CLINICAL TRIAL: NCT01824628
Title: Comparaison Des Intervalles QT/QTc Entre Une Population HIV Positive Ambulatoire Sous thérapie antirétrovirale et Une Population Ambulatoire HIV négative
Brief Title: Comparison of the QT/QTc Interval Between an Outpatient HIV-Infected Population on Antiretroviral Therapy and Two Large HIV-Negative Cohorts
Acronym: QTVIE
Status: Completed | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Other Study IDs: CE12.316
Record Dates: First submitted 2013-04-02; First posted 2013-04-05 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: QT and Corrected QT Intervals Prolongation in HIV Positive Subjects Treated With an Antiretroviral Regimen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 10 mL whole blood in a purple Vacutainer EDTA tube
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- • HIV positive subjects receiving antiretroviral regimen
- • HIV negative subjects from the pre-admission surgical clinic

SUMMARY:
This is a unicentric, two cohorts, observational transversal study.

The purpose of this study is to compare the QT/QTc intervals of HIV positive subjects receiving an antiretroviral therapy and those without HIV in an ambulatory care setting.

DETAILED DESCRIPTION:
Primary objective:

The primary objective is to compare the QT/QTc intervals of HIV positive subjects treated with antiretroviral therapy and followed at the ambulatory HIV clinic and the QT/QTc intervals of :

1. an outpatient HIV negative population from the same health center pre-admission one-day surgical clinic.
2. the large HIV-free korean population studied in the ECG-ViEW database.

Secondary objectives :

* Evaluate the prevalence of QTc interval prolongation in the outpatient HIV positive population comparatively to the two HIV negative outpatient populations available from the one-day surgical clinic and the ECG-ViEW database.
* Evaluate risk factors associated with QTc interval prolongation in the outpatient HIV positive population compared to the outpatient HIV negative population and the population studied in the ECG-ViEW database.
* Compare the QT/QTc intervals and the prevalence of QTc interval prolongation of the outpatient HIV positive population currently on an antiretroviral regimen including a protease inhibitor versus those on an antiretroviral regimen without protease inhibitor.
* Compare the QT/QTc intervals among the outpatient HIV positive population treated with a protease inhibitor, in regard to the presence or the absence of certain genetic polymorphisms that may influence pharmacokinetic aspects of protease inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Age eligible for study : 18-65 years old inclusively
* Gender eligible for study : Both

Exclusion Criteria:

* Hospitalised at the moment of recruitment
* AIDS status

  o Opportunistic infections acquired in the last 30 days before the date of recruitment
* Age < 18 years old and > 65 years old
* Follow-up care in an oncology clinic
* Dialysis during the study period
* Pregnancy
* Without antiretroviral therapy
* History of a myocardial infarction in the 3 weeks preceding recruitment
* Have a pacemaker
* Diagnosed with bundle branch block on ECG
* Principal follow-up care outside of the CHUM HIV clinic
* Refusal to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study is being conducted within the Centre hospitalier de l'Université de Montréal (CHUM). The recruited population was identified from the CHUM ambulatory care HIV clinic and an ECG registry composed of outpatient HIV negative subjects who were scheduled for a one-day surgery. The HIV positive outpatients on antiretroviral therapy will be recruited prospectively from March 2013 through August 2013. The outpatient HIV negative cohort will be recruited retrospectively according to a 10:1 ratio.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2013-03; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
QT and corrected QT (QTc) intervals determined by a 12-leads ECG | Day 0 = Day 1 - This is a transversal study.
  The QT/QTc intervals are determined by a 50 mm/s 12-leads ECG in the outpatient HIV positive population. The ECG is conducted in the morning, between 8:00 and 12:00 to limit the circadian variation.
  For the control group, the QT/QTc intervals are assessed through a registry of outpatient HIV negative subjects who had had a standard 12-leads ECG done in pre-admission one-day surgery clinic.
  In both groups, the corrected QT interval is calculated with the Bazett's formula and the Fridericia's formula.

SECONDARY OUTCOMES:
Prevalence of QTc interval prolongation in both study groups | Day 0 = Day 1 - This is a transversal study.
  Compare the QTc intervals calculated with the Bazett's formula and the Fridericia's formula in both study groups in order to determine the prevalence of QTc interval prolongation. The QTc interval is considered to be prolonged if it exceeds 430 ms in women and 450 ms in men.
To assess risk factors of QTc interval prolongation in both study groups | Day 0 = Day 1 - This is a transversal study.
  A predetermined questionnaire is filled for each of the study subjects in order to assess factors associated with an increased QTc interval prolongation. This contains demographic information (age, sex, ethnicity...), known health issues (cardiovascular diseases, diabetes, liver diseases...), concomitant drugs, etc.
Prevalence of QT/QTc intervals prolongation and associated risk factors among outpatient HIV subjects | Day 0 = Day 1 - This is a transversal study.
  Compare the QTc intervals calculated with the Bazett's formula and the Fridericia's formula between outpatient HIV positive subjects treated with a protease inhibitor (PI) based antiretroviral regimen and those treated with an antiretroviral regimen without PI. The QTc interval is considered to be prolonged if it exceeds 430 ms in women and 450 ms in men.
Evaluate the influence of genetic polymorphisms on PI's pharmacokinetic metabolisms in outpatient HIV positive subjects treated with a PI | Day 0 = Day 1 - This is a transversal study
  A blood sample of each subject treated with a PI is analyzed in the laboratory in order to determine whether certain genetic polymorphisms influence on the metabolism of the drug, thus causing a QTc interval prolongation or not.

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Turgeon, B. Pharm., M. Sc., Ph. D., Principal Investigator — Centre de Recherche du Centre Hospitalier de l'Université de Montréal
Locations (1):
- Unité Hospitalière de Recherche et d'Enseignement et de Soins sur le Sida (UHRESS) ; Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada